CLINICAL TRIAL: NCT06994416
Title: A Novel Fluorescent Ductal Needle With Controllable Detachment for Real-time Localization and Sampling of High-risk Breast Micro Lesions: a Retrospective Study
Brief Title: A Novel Fluorescent Ductal Needle for Localization and Sampling of High-risk Breast Micro Lesions
Status: Recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, JIAN WEN, Deputy Director of the Fifth General Surgery Department, The Fourth Affiliated Hospital of China Medical University
Other Study IDs: FourthAHChinaMU
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Mammary Tumor; Nipple Discharge
Keywords: micro lesions; breast duct; fluorescent ductal needle; localization needle; controllable detachment
MeSH Terms: conditions — Breast Neoplasms; Galactorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Patients received breast ductal excision surgery utilizing a novel fluorescent localization marker needle. Specimens were submitted for intraoperative frozen section analysis as well as for postoperative paraffin-embedded pathological evaluation.
  Interventions: Device: novel fluorescent localization marker needle
- Control: Patients received breast ductal excision surgery utilizing conventional localization methods. Specimens were submitted for intraoperative frozen section analysis as well as for postoperative paraffin-embedded pathological evaluation.
  Interventions: Device: conventional localization marker needle

INTERVENTIONS:
Device: novel fluorescent localization marker needle — novel fluorescent localization needle, which features a controllable shedding quantum dot chiral nanofluorescent coating
  Groups: Experimental
Device: conventional localization marker needle — conventional localization marker needle, without any coating
  Groups: Control

SUMMARY:
This retrospective cohort study investigates the differences in the reliability of rapid pathology compared to postoperative pathology when utilizing a novel fluorescent localization needle equipped with a controllable shedding quantum dot chiral nanofluorescent coating, in contrast to traditional localization techniques for breast duct lesions. The primary goal is to evaluate the clinical effectiveness of this innovative fluorescent localization needle in facilitating accurate pathological diagnoses of micro lesions situated within breast ducts.

DETAILED DESCRIPTION:
The diameter of breast ducts is less than 0.7 mm, which poses a considerable technical challenge in the accurate localization of early-stage small lesions during surgical and pathological sampling. These early micro lesions typically measure on the millimeter scale, necessitating an increased excision margin by surgeons to reduce the risk of overlooking them. However, this practice complicates the pathologists' ability to accurately identify these micro lesions during diagnosis, thereby heightening the likelihood of missed diagnoses and the potential for additional surgeries for patients. Current localization methods, such as liquid methylene blue and traditional localization needles, demonstrate a high rate of pathological missed diagnoses due to inaccuracies in localization and specimen contamination. Therefore, there is an urgent need for the development of innovative localization technologies that can facilitate the precise identification of millimeter-scale micro lesions within breast ducts and improve the accuracy of pathological sampling. This study aims to conduct a retrospective analysis to compare the consistency of intraoperative and postoperative pathological assessments between a novel fluorescent localization needle, which features a controllable shedding quantum dot chiral nanofluorescent coating, and conventional localization techniques used during breast duct lesion surgeries. The objective is to evaluate the clinical utility of the new fluorescent localization needle in the accurate pathological diagnosis of micro lesions within breast ducts and to enhance the precision of pathological assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years.
2. Patients who have been diagnosed intraductal breast lesion by ductoscopy.
3. Patients who have undergone ductal excision.
4. Patients who are capable of providing written informed consent and adhering to the study protocols.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Patients who have known allergy to quantum-dot materials or localization needle components.
3. Patients with active hepatitis B or C infection with detectable viral load.
4. Patients with unstable cardiovascular disease (e.g., recent myocardial infarction, uncontrolled arrhythmia, NYHA class III-IV heart failure).
5. Patients with history of neurological or psychiatric disorders that may impair compliance (e.g., epilepsy, dementia).
6. Patients who concurrent participation in another interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study estimated enroll 300 patients diagnosed with intraductal breast lesion by ductoscopy at the Fourth Affiliated Hospital of China Medical University between January 2023 and December 2024. All participants met inclusion criteria, and underwent ductal excision utilizing a novel fluorescent localization marker needle or conventional localization methods.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
pathological assessment concordance rates | Data analysis period: June 2025- December 2025
  Evaluate and compare the discrepancies in the consistency of intraoperative frozen and postoperative paraffin-embedded pathological assessments between subjects undergoing breast duct excision surgery utilizing a novel fluorescent localization marker needle and those employing conventional localization methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wen, MD, Principal Investigator — The Fourth Affiliated Hospital of China Medical University
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alshurbasi N, Cartlidge CWJ, Kohlhardt SR, Hadad SM. Predicting Patients Found to Have Malignancy at Nipple Duct Surgery. Breast Care (Basel). 2020 Oct;15(5):491-497. doi: 10.1159/000504528. Epub 2019 Dec 13. PMID 33223992